CLINICAL TRIAL: NCT03723824
Title: An Open-label, Cohort Study of Grazoprevir/Elbasvir Combination Therapy for Patients With Genotype 1b Chronic Hepatitis C After Liver or Kidney Transplantation
Brief Title: Grazoprevir/Elbasvir for Genotype 1b Chronic Hepatitis C After Liver or Kidney Transplantation
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: COV-19 pandemic
Sponsor: Taichung Veterans General Hospital (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Teng-Yu Lee, Principle Investigator of the Liver Disease Center, Taichung Veterans General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SF18281A
Record Dates: First submitted 2018-10-26; First posted 2018-10-30 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Chronic Hepatitis c; Liver Transplant Infection; Kidney Transplant Infection
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — grazoprevir; elbasvir; elbasvir-grazoprevir drug combination

STUDY DESIGN:
Intervention Model Description: grazoprevir 100 mg/ elbasvir 50 mg, Zepatier®, 1# qd for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Zepatier therapy (Experimental): grazoprevir 100 mg/ elbasvir 50 mg (Zepatier®, MSD) once daily for 12 weeks
  Interventions: Drug: grazoprevir 100 mg/ elbasvir 50 mg, Zepatier®

INTERVENTIONS:
Drug: grazoprevir 100 mg/ elbasvir 50 mg, Zepatier® — grazoprevir 100 mg/ elbasvir 50 mg (Zepatier®, MSD) once daily for 12 weeks
  Other Names: Zepatier

SUMMARY:
Grazoprevir/elbasvir combination therapy is highly effective in the treatment of genotype 1b chronic hepatitis C, and the drug-drug interaction with central immunosuppressant, such as tacrolimus, should be manageable. The aim of this study is to assess the efficacy and tolerability of grazoprevir/elbasvir combination therapy in treating genotype 1b chronic hepatitis C after liver or kidney transplantation.

DETAILED DESCRIPTION:
Grazoprevir/elbasvir combination therapy (grazoprevir 100 mg/ elbasvir 50 mg, Zepatier®, MSD) has been recommended as the 1st-line treatment for genotype 1b chronic hepatitis C by the updated international guidelines, and the rates of sustained virologic response (SVR) can be higher than 95% in either treatment-naïve or peginterferon-experienced patients with genotype 1b chronic hepatitis C. Moreover, even among patients with liver cirrhosis, the efficacy of grazoprevir/elbasvir combination therapy remains very high. In addition, drug-related adverse effects (AEs) were quite low in previous studies, and less than 1% of cirrhotic patients discontinued this therapy during treatment period (4). Grazoprevir/elbasvir combination therapy is an effective and safe treatment for chronic hepatitis C.

Chronic hepatitis C is one of the most common indications for liver transplantation. Patients underwent liver or kidney transplantation always suffer from recurrent chronic hepatitis C. Recurrent chronic hepatitis C can result in liver cirrhosis, liver decompensation, and death. Chronic hepatitis C is also associated with a higher incidence of chronic rejection, graft failure and mortality after kidney transplantation. Treating hepatitis C virus (HCV) infection after liver or kidney transplantation was a big challenge before the development of new direct-acting antiviral (DAA). Not only a low SVR rate but also a high rate of severe adverse effects results in the hesitation of peginterferon-ribavirin combination therapy. Although some new DAAs can be used in organ transplantation, the cost remains quite high. More new DAA choices for patients underwent organ transplantation are needed.

The clinical data of grazoprevir/elbasvir combination therapy on the treatment for patients with chronic hepatitis C after liver or kidney transplantation remain lacking. With high virologic response rates and low adverse effects in the management for chronic hepatitis C, grazoprevir/elbasvir combination therapy could be a good option for patients underwent liver or kidney transplantation. No drug-drug interaction (DDI) was noted between grazoprevir/elbasvir combination therapy and steroid, and the DDI with the most commonly-used immunosuppressant, tacrolimus, was also not significant, The drug levels of immunosuppressants can be carefully monitored and adjusted during treatment period. The aim of this study is to assess the efficacy and tolerability of grazoprevir/elbasvir combination therapy in treating genotype 1b chronic hepatitis C after liver or kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. At least 20 years of age
2. Chronically infected with genotypes 1b HCV
3. Underwent liver and/ or kidney transplantation
4. Without clinical or pathologic evidence of moderate or severe rejection

Exclusion Criteria:

1. HCV genotype other than 1b
2. Liver decompensation (Child-Pugh score > 6)
3. Co-infected with human immunodeficiency virus: Positive HIV1/2 or hepatitis B virus : Positive HBsAg and detected HBV DNA
4. Prior exposure to an NS5A inhibitor
5. Any active malignancies
6. Hemoglobin level less than 10 g/dl
7. Platelet level of 75,000/mm3 or less
8. Alanine aminotransferase, aspartate aminotransferase, or alkaline phosphatase level 10 times or more the upper limit of normal
9. Total bilirubin level greater than 3 times or more the upper limit of normal
10. Albumin less than 3 g/dL
11. Using medication that is not considered safe to co-administer with , such as cyclosporine
12. Pregnant or breast-feeding women
13. Known allergy to grazoprevir or elbasvir

(Unregistered liver or kidney transplant in other countries is illegal in Taiwan)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2021-03-13 (Actual)

PRIMARY OUTCOMES:
Sustained virologic response (SVR) | At post-treatment week 12
  The HCV viral load (IU/mL) in blood at post-treatment week 12 (SVR12)

SECONDARY OUTCOMES:
Adverse effects (AEs) | During the treatment period (the 1st, 2nd, 4th, 6th, 8th, 10th, 12th weeks)
  Any AEs during the treatment period
Used immunosuppressant blood levels | During the treatment period (the 1st, 2nd, 4th, 6th, 8th, 10th, 12th weeks)
  The immunosuppressant concentration (ng/mL) in blood during the treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Teng-Yu Lee, MD, Principal Investigator — Taichung Veterans General Hospital
Locations (2):
- Taiwan (2):
  - Taichung Veterans General Hospital, Taichung
  - China Medical University Hospital, Taichung

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zeuzem S, Ghalib R, Reddy KR, Pockros PJ, Ben Ari Z, Zhao Y, Brown DD, Wan S, DiNubile MJ, Nguyen BY, Robertson MN, Wahl J, Barr E, Butterton JR. Grazoprevir-Elbasvir Combination Therapy for Treatment-Naive Cirrhotic and Noncirrhotic Patients With Chronic Hepatitis C Virus Genotype 1, 4, or 6 Infection: A Randomized Trial. Ann Intern Med. 2015 Jul 7;163(1):1-13. doi: 10.7326/M15-0785. PMID 25909356
- [Result] Kwo P, Gane EJ, Peng CY, Pearlman B, Vierling JM, Serfaty L, Buti M, Shafran S, Stryszak P, Lin L, Gress J, Black S, Dutko FJ, Robertson M, Wahl J, Lupinacci L, Barr E, Haber B. Effectiveness of Elbasvir and Grazoprevir Combination, With or Without Ribavirin, for Treatment-Experienced Patients With Chronic Hepatitis C Infection. Gastroenterology. 2017 Jan;152(1):164-175.e4. doi: 10.1053/j.gastro.2016.09.045. Epub 2016 Oct 5. PMID 27720838
- [Result] Jacobson IM, Lawitz E, Kwo PY, Hezode C, Peng CY, Howe AYM, Hwang P, Wahl J, Robertson M, Barr E, Haber BA. Safety and Efficacy of Elbasvir/Grazoprevir in Patients With Hepatitis C Virus Infection and Compensated Cirrhosis: An Integrated Analysis. Gastroenterology. 2017 May;152(6):1372-1382.e2. doi: 10.1053/j.gastro.2017.01.050. Epub 2017 Feb 11. PMID 28193518
- [Derived] Lai PC, Chen CH, Jeng LB, Yu TM, Tsai SF, Wu MJ, Cheng SB, Yang SS, Lee TY. Grazoprevir/Elbasvir Treatment in Liver or Kidney Transplant Recipients with Genotype 1b Hepatitis C Virus Infection. Antimicrob Agents Chemother. 2022 Feb 15;66(2):e0200321. doi: 10.1128/AAC.02003-21. Epub 2021 Dec 13. PMID 34902265